CLINICAL TRIAL: NCT00493272
Title: Fibrinogen vs Placebo for Improvement of Clot Strength
Brief Title: Dilutional Coagulopathy in Patients Undergoing Elective Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Christian Fenger-Eriksen (Other)
Responsible Party: Sponsor-Investigator, Christian Fenger-Eriksen, PhD MD, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20070037
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Blood Coagulation Disorder
Keywords: Blood coagulation disorder, acquired; Hemodilution; Fibrinogen; Hemostasis; HES
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Fibrinogen; Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Nacl
  Interventions: Drug: Fibrinogen
- Fibrinogen (Active Comparator): Fibrinogen
  Interventions: Drug: Fibrinogen

INTERVENTIONS:
Drug: Fibrinogen — Fibrinogen behandling
  Other Names: Active drug

SUMMARY:
The purpose of the present study is to perform a comprehensive description of haemostasis parameters before and after haemodilution with Hydroxyethyl starch (HES) following acute bleeding during elective surgery. Moreover the study aims to test the in vivo haemostatic potential of fibrinogen concentrate in dilutional coagulopathy caused by HES in a clinical, prospective, placebo-controlled randomised setup.

We hypothesise; a) A coagulopathy is induced following in vivo haemodilution; b) the coagulopathy is improved or partially improved by fibrinogen.

DETAILED DESCRIPTION:
Background Hydroxyethyl starch (HES) is a group of artificial colloid solutions widely used for plasma expansion and volume resuscitation. HES consist of branched chains of hydroxylated glucose molecules defined by average molecular weight, degree of hydroxyethylation, and C2/C6 ratio. Several clinical reports and in vitro experiments have documented an impaired coagulation system induced by haemodilution with HES and other colloid plasma expanders. The exact mechanisms responsible for HES induced coagulopahty are not fully understood although reduced levels of von Willebrand factor (vWF), acquired platelet dysfunction, reduced factor VIII levels, and dysfunctional fibrinogen polymerization seems to reflect an important aspect of the pathogenesis.

Experimental laboratory studies performed in our centre and verified by several other research groups have shown successful reversal of the colloid plasma expander induced coagulopathy by fibrinogen concentrate.10-13 So far, the present knowledge are based on laboratory experiments and animal studies. Hence, it appears desirable to perform a comprehensive description of haemostasis parameters following HES induced dilutional coagulopathy in an acute clinical bleeding situation.

Materials and Methods

Study design: Clinical, prospective, double-blind, randomised, place-controlled trial. Blood samples:

Primary end point:

Dynamic whole blood clot formation

Secondary end points:

A) Single coagulation factor activities B) Platelet function C) Whole blood clot stability. D) Thrombin generation

Perspectives:

Serious surgical and traumatic bleedings are common and associated with a high mortality rate. The present study can significantly contribute to our overall understanding of the mechanisms involved in HES induced dilutional coagulopathy.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Indication for performing cystectomia
* Written informed consent

Exclusion Criteria:

* Uses of acetyl-salicylic or non-steroid anti-inflammatory drugs 2 days prior to blood sampling.
* Abnormal preoperative coagulations parameters (Platelets, PP, APTT, D- dimer, Fibrinogen, AT, TT)
* Disseminated cancer and/or bone metastasis
* Medical history of ischemic heart disease, claudicatio, or arteriosclerosis
* Medical history of previous thrombo-embolic event
* Renal failure defined as clinical relevant abnormal levels of creatinine
* Liver failure defined as clinical relevant abnormal levels of ALAT
* Hypersensibility to Voluven, Haemocomplettan or ingredients
* Fertile women not using safe contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Dynamic whole blood clot formation. | 60 minutes

SECONDARY OUTCOMES:
A) Single coagulation factor activities B) Platelet function C) Whole blood clot stability. D) Thrombin generation. | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Else Tønnesen, MD, Prof, Principal Investigator — Aarhus University Hospital, Department of Anaesthesiology
Locations (1):
- Aarhus University Hospital, Department of Anaesthesiology, Dk-8200 Aarhus N, Denmark

REFERENCES:
- [Background] Jamnicki M, Zollinger A, Seifert B, Popovic D, Pasch T, Spahn DR. Compromised blood coagulation: an in vitro comparison of hydroxyethyl starch 130/0.4 and hydroxyethyl starch 200/0.5 using thrombelastography. Anesth Analg. 1998 Nov;87(5):989-93. doi: 10.1097/00000539-199811000-00002. PMID 9806670
- [Background] Damon L, Adams M, Stricker RB, Ries C. Intracranial bleeding during treatment with hydroxyethyl starch. N Engl J Med. 1987 Oct 8;317(15):964-5. doi: 10.1056/NEJM198710083171517. No abstract available. PMID 2442613
- [Background] Baldassarre S, Vincent JL. Coagulopathy induced by hydroxyethyl starch. Anesth Analg. 1997 Feb;84(2):451-3. doi: 10.1097/00000539-199702000-00040. No abstract available. PMID 9024047
- [Background] de Jonge E, Levi M, Buller HR, Berends F, Kesecioglu J. Decreased circulating levels of von Willebrand factor after intravenous administration of a rapidly degradable hydroxyethyl starch (HES 200/0.5/6) in healthy human subjects. Intensive Care Med. 2001 Nov;27(11):1825-9. doi: 10.1007/s001340101107. Epub 2001 Sep 26. PMID 11810130
- [Background] Fenger-Eriksen C, Anker-Moller E, Heslop J, Ingerslev J, Sorensen B. Thrombelastographic whole blood clot formation after ex vivo addition of plasma substitutes: improvements of the induced coagulopathy with fibrinogen concentrate. Br J Anaesth. 2005 Mar;94(3):324-9. doi: 10.1093/bja/aei052. Epub 2004 Dec 17. PMID 15608046
- [Background] Fenger-Eriksen C, Ingerslev J, Sorensen B. Coagulopathy induced by colloid plasma expanders--search for an efficacious haemostatic intervention. Acta Anaesthesiol Scand. 2006 Aug;50(7):899-900. doi: 10.1111/j.1399-6576.2006.01054.x. No abstract available. PMID 16879481